CLINICAL TRIAL: NCT05439356
Title: Colchicine in High-risk Patients With Acute Minor-to-moderate Ischemic Stroke or Transient Ischemic Attack (CHANCE-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCRC-2022-05
Record Dates: First submitted 2022-06-20; First posted 2022-06-30 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke; TIA
MeSH Terms: conditions — Ischemic Stroke | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine Group (Experimental): Patients in this arm will receive colchicine for 90 days in addition to standard medical care
  Interventions: Drug: Colchicine
- Placebo Colchicine Group (Placebo Comparator): Patients in this arm will receive placebo colchicine for 90 days in addition to standard medical care
  Interventions: Drug: Placebo colchicine

INTERVENTIONS:
Drug: Colchicine — Oral colchicine will be initiated with a dose of 1mg per day (one tablet of 0.5mg initially followed by another tablet of 0.5 mg at least four hours later) on days 1 through 3, and continuing with 0.5 mg (one tablet) per day on days 4 through 90.
  Arms: Colchicine Group
Drug: Placebo colchicine — Oral placebo colchicine will be initiated with a dose of 1mg per day (one tablet of 0.5mg initially followed by another tablet of 0.5 mg at least four hours later) on days 1 through 3, and continuing with 0.5 mg (one tablet) per day on days 4 through 90.
  Arms: Placebo Colchicine Group

SUMMARY:
This study is a multicentre, randomized, double-blind, placebo-controlled, investigator-sponsored study that aims to investigate the efficacy of colchicine in preventing recurrent stroke in the patients with acute minor-to-moderate ischemic stroke or TIA and a hsCRP level of ≥2mg/L.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled trial that aims to investigate the efficacy of colchicine in preventing recurrent stroke in the patients with acute minor-to-moderate ischemic stroke or TIA and a hsCRP level of ≥2mg/L. Patients who were eligible to the inclusion criteria and ineligible to the exclusion criteria will be randomly assigned into two groups by a 1:1 ratio. Patients in one arm will receive colchicine initiated with a dose of 1mg per day on days 1 through 3, and continuing with 0.5 mg per day on days 4 through 90, and those in the other arm will receive an equivalent placebo drug. Study visits will be performed on the day of randomization, at discharge, at day 90 and at 1 year. The primary outcome was stroke (ischemic or hemorrhagic) during 90 days of follow-up in an intention-to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years or older than 40 years；
2. Acute cerebral ischemic event due to： Acute minor-to-moderate ischemic stroke (NIHSS≤5 at the time of randomization) or TIA with moderate-to-high risk of stroke (ABCD2 score ≥ 4 at the time of randomization)；
3. With a hsCRP level of ≥2mg/L at randomization;
4. Can be treated with study drug within 24 hours of symptoms onset*(*Symptom onset is defined by the "last seen normal" principle)；
5. Informed consent signed.

Exclusion Criteria:

1. Malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head CT or MRI.
2. Isolated or pure sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI.
3. Iatrogenic causes (angioplasty or surgery) of stroke or TIA.
4. Presumed cardiac source of embolus, such as atrial fibrillation or prosthetic cardiac valve).
5. A score of ≥ 2 on the modified Rankin scale immediately before the occurrence of the index event.
6. Usage of colchicine within 30 days before randomization or planning to take colchicine therapy for other indications.
7. Known allergy or sensitivity or intolerance to colchicine.
8. Inflammatory bowel disease (Crohn's or ulcerative colitis) or chronic diarrhea.
9. Symptomatic peripheral neuropathy or pre-existing progressive neuromuscular disease or with creatine kinase (CK) level > 3 times the upper limit of normal as measured within the past 30 days and determined to be non-transient through repeat testing.
10. A history of cirrhosis, chronic active hepatitis or severe hepatic disease.
11. Impaired hepatic (ALT or AST > twice the upper limit of normal range) or kidney (creatinine exceeding 1.5 times of the upper limit of normal range or eGFR less than 50 ml/min) function at randomization.
12. Anemia (haemoglobin <10g/dL), thrombocytopenia (platelet count <100×109/L) or leucopenia (white blood cell <3×109/L) at randomization.
13. In the acute phase of respiratory tract infection, urinary tract infection, and gastro-enteritis, or currently using or planning to receive oral or intravenous anti-infective therapy for any other infection.
14. Currently using or planning to begin long-term (>7 days) systemic anti-inflammatory drugs (NSAIDs except for aspirin, oral or intravenous steroid therapy) during the study.
15. Planning to use moderate or strong CYP3A4 inhibitors (clarithromycin, erythromycin, telithromycin, other macrolide antibiotics, ketoconazole, itraconazole, voriconazole, ritonavir, atazanavir, indinavir, other HIV protease inhibitors, verapamil, diltiazem, quinidine, digoxin, disulfiram, etc) or P-gp inhibitors (cyclosporine) at randomization.
16. Planned surgery or interventional treatment requiring cessation of the study drug during the study.
17. Participating in another clinical trial with an investigational drug or device concurrently or during the last 30 days.
18. Women of childbearing age who were not practicing reliable contraception and did not have a documented negative pregnancy test or severe noncardiovascular coexisting condition.
19. Severe non-cardiovascular comorbidity with a life expectancy of less than 3 months.
20. With a history of clinically significant drug or alcohol abuse.
21. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders, or to be an unsuitable candidate for the study for any other considered by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8343 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Any new stroke events | any time within 90 days
  Incidence of any new ischemic or hemorrhagic stroke

SECONDARY OUTCOMES:
New vascular events | any time within 90 days
  Incidence of any new vascular events, including ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular death
New ischemic stroke | any time within 90 days
  Incidence of any new ischemic stroke
Poor functional outcome | at 90 days after randomization
  Rate of poor functional outcome defined as a Modified Rankin Scale score of >1 (Modified Rankin Scale score ranges from 0 (no symptoms) to 6 (death) and higher score means worse outcome)
New stroke and TIA | any time within 90 days
  Incidence of any new stroke and TIA
Severity of recurrent stroke and TIA | within 90 days after randomization
  Severity is measured using a six-level ordered categorical scale that incorporates the mRS: fatal stroke [mRS 6]/severe non-fatal stroke [mRS 4 or 5]/moderate stroke [mRS 2 or 3]/mild stroke [mRS 0 or 1]/TIA/no stroke-TIA

OTHER OUTCOMES:
Any new stroke events | any time within 1 year after randomization
  Incidence of any new ischemic or hemorrhagic stroke
New vascular events | any time within 1 year after randomization
  Incidence of any new vascular events, including ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular death
New ischemic stroke | any time within 1 year after randomization
  Incidence of any new ischemic stroke
Poor functional outcome | at 1 year after randomization
  Rate of poor functional outcome defined as a Modified Rankin Scale score of >1 (Modified Rankin Scale score ranges from 0 (no symptoms) to 6 (death) and higher score means worse outcome)
New stroke and TIA | any time within 1 year after randomization
  Incidence of any new stroke and TIA
Severity of recurrent stroke and TIA | within 1 year after randomization
  Severity is measured using a six-level ordered categorical scale that incorporates the mRS: fatal stroke [mRS 6]/severe non-fatal stroke [mRS 4 or 5]/moderate stroke [mRS 2 or 3]/mild stroke [mRS 0 or 1]/TIA/no stroke-TIA
Adverse events | within 90 days
  Rate of adverse events ( AEs )
Severe adverse events | within 90 days
  Rate of serious adverse events ( SAEs )
Increased CK levels or abnormal hepatic function when concomitant high-intensity statin treatment | within 90 days
  Rate of increased CK levels (≥ 5 times the upper limit of normal) or abnormal hepatic function (ALT or AST ≥ 3 times the upper limit of normal range) within 90 days when concomitant high-intensity statin treatment
Adverse events | within 1 year
  Rate of adverse events ( AEs )
Severe adverse events | within 1 year
  Rate of serious adverse events ( SAEs )

CONTACTS AND LOCATIONS:
Locations (244):
- China (244):
  - Linquan County People's Hospital, Fuyang, Anhui
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The First People's Hospital of Wuhu, Wuhu, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shunyi Airport Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Fuxing Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing, Beijing Municipality
  - Chongqing Sanbo Chang 'an Hospital, Chongqing, Chongqing Municipality
  - Chongqing Tungwah Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Fuling Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical and Pharmaceutical College, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xiushan Tujia and Miao Autonomous County People's Hospital, Chongqing, Chongqing Municipality
  - Ningde People's Hospital, Ningde, Fujian
  - The Sanming First Hospital Affiliated to Fujian Medical University, Sanming, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - The Third Hospital of Xiamen, Xiamen, Fujian
  - The First People's Hospital of Lanzhou City, Lanzhou, Gansu
  - Zhangye People's Hospital Affiliated To Hexi University, Zhangye, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong second Provincial Central Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Jinan University (Heyuan Shenhe People's Hospital), Heyuan, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - Baise City People's Hospital, Baise City, Guangxi
  - The People's Hospital of Cenxi City, Wuzhou, Guangxi
  - Guihang Guiyang hospital, Guizhou, Guiyang
  - Puding County People's Hospital, Anshun, Guizhou
  - Zhejiang Provincial People's Hospital Bijie Hospital, Bijie, Guizhou
  - The First People's Hospital of Guiyang, Guiyang, Guizhou
  - The Second People's Hospital of Guiyang, Guiyang, Guizhou
  - The Third People's Hospital of Guiyang, Guiyang, Guizhou
  - The People's Hospital of the Qiandongnan Miao and Dong Autonomous Prefecture, Kaili, Guizhou
  - The second Affiliated Hospital of Guizhou Medical University, Kaili, Guizhou
  - Qianxinan Buyi and Miao Autonomous Prefecture People's Hospital, Xingyi, Guizhou
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Baoding Xushui District People's Hospital, Baoding, Hebei
  - Hebei Tang County People Hospital, Baoding, Hebei
  - Shunping County Hospital, Baoding, Hebei
  - The Hospital of Anguo City, Baoding, Hebei
  - Wangdu County Hospital,Hebei Province, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Chengde County Hospital, Chengde, Hebei
  - Guantao county central Hospital, Handan, Hebei
  - Handan First Hospital, Handan, Hebei
  - Qiu County Hospital of Traditional Chinese Medicine, Handan, Hebei
  - Qiu County People's Hospital, Handan, Hebei
  - Hejian People's Hospital, Hejian, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - The No.4 People's Hospital of Hengshui(Department of Neurology ward 1), Hengshui, Hebei
  - The No.4 People's Hospital of Hengshui(Department of Neurology ward 2), Hengshui, Hebei
  - Shijiazhuang Third Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University of Science And Technology Affiliated Hospital, Tangshan, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Qinghe people's hospital, Xingtai, Hebei
  - Werixian People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hongxinglong Hospital of Beidahuang Group, Shuangyashan, Heilongjiang
  - The People's Hospital of Anyang City, Anyang, Henan
  - Dengzhou Central Hospital, Dezhou, Henan
  - Hebi Coal Industry (Group) Co., Ltd. General Hospital, Hebi, Henan
  - Boai People's Hospital, Jiaozuo, Henan
  - Mengzhou Hospital of Traditional Chinese Medicine, Jiaozuo, Henan
  - Mengzhou People's Hospital(Department of Neurology ward 1), Jiaozuo, Henan
  - Mengzhou People's Hospital(Department of Neurology ward 2), Jiaozuo, Henan
  - Qinyang City Hospital of Traditional Chinese Medicine, Jiaozuo, Henan
  - Qinyang People's Hospital, Jiaozuo, Henan
  - Wuzhi County People's Hospital, Jiaozuo, Henan
  - Xiuwu County People's Hospital, Jiaozuo, Henan
  - Jiyuan Hospital of Traditional Chinese Medicine, Jiyuan, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Lankao County Central Hospital, Kaifeng, Henan
  - Weishi Central Hospital, Kaifeng, Henan
  - Luoning County People's Hospital, Luoyang, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Luoyang Dongfang People's Hospital, Luoyang, Henan
  - Luoyang First People's Hospital, Luoyang, Henan
  - Luoyang Mengjin District People's Hospital, Luoyang, Henan
  - Ruyang People's Hospital, Luoyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Yiyang County People's Hospital, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - Neixiang County People's Hospital, Nanyang, Henan
  - Xichuan County People's Hospital, Nanyang, Henan
  - Xixia County People's Hospital, Nanyang, Henan
  - Ruzhou People's Hospital, Pingdingshan, Henan
  - The second people's hospital of Pingdingshan, Pingdingshan, Henan
  - Ye County People's Hospital, Pingdingshan, Henan
  - Fanxian People's Hospital, Puyang, Henan
  - Puyang County People's Hospital, Puyang, Henan
  - Qingfeng xinxing hospital, Puyang, Henan
  - The First People Hospital of Lingbao, Sanmenxia, Henan
  - Sui county traditional Chinese medicine hospital, Shangqiu, Henan
  - The Fourth People's Hospital of Shangqiu, Shangqiu, Henan
  - The Shangqiu First People's Hospital, Shangqiu, Henan
  - Zhecheng People's Hospital, Shangqiu, Henan
  - Huixian People's Hospital, Xinxiang, Henan
  - The second People Hospital of Xinxiang Henan, Xinxiang, Henan
  - Xinxiang tongmeng hospital, Xinxiang, Henan
  - The Affiliated Hospital of Xinyang Vocational and Technical College, Xinyang, Henan
  - Central Hospital of Yongcheng, Yongcheng, Henan
  - Xingyang People's Hospital, Zhengzhou, Henan
  - Xinmi Hospital of T.C.M, Zhengzhou, Henan
  - Shenqiu County People's Hospital, Zhoukou, Henan
  - Taikang Xian People's Hospital, Zhoukou, Henan
  - Xihua Xian People's Hospital, Zhoukou, Henan
  - Zhumadian TCM Hospital, Zhumadian, Henan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hunan
  - The Fourth People's Hospital of Chenzhou, Chenzhou, Hunan
  - The Third People's Hospital of Chenzhou, Chenzhou, Hunan
  - Hengyang Central Hospital, Hengyang, Hunan
  - Shaodong People's Hospital, Shaoyang, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Baotou City Central Hospital, Baotou, Inner Mongolia
  - Sinopharm North Hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The people's Hospital of Wulateqianqi, Bayan Nur, Inner Mongolia
  - Wuyuan County People's Hospital, Bayan Nur, Inner Mongolia
  - Huhhot First Hospital, Hohhot, Inner Mongolia
  - Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Inner Mongolia Forestry General Hospital, Hulunbuir, Inner Mongolia
  - Ordos central hospital, Ordos, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Minzu University, Tongliao, Inner Mongolia
  - Tongliao City Hospital, Tongliao, Inner Mongolia
  - Ulanpab Central Hospital, Ulanqab, Inner Mongolia
  - The people's Hospital of Wuhai, Wuhai, Inner Mongolia
  - Tuoketuo County Hospital, Hohhot, Inner Mongoria
  - Nanjing Gaochun People's Hospital, Nanjing, Jiangsu
  - Jiangsu Rudong County People's Hospital, Nantong, Jiangsu
  - Nantong Tongzhou District No.8 People's Hospital, Nantong, Jiangsu
  - Suxitong Science and Technology Industrial Park People's Hospital, Nantong, Jiangsu
  - The People's Hospital of Rugao, Nantong, Jiangsu
  - The Sixth People's Hospital of Nantong, Nantong, Jiangsu
  - Nanjing Drum Tower Hospital Group Suqian Hospital, Suqian, Jiangsu
  - Siyang kangda hospital, Suqian, Jiangsu
  - Xinghua City People's Hospital, Taizhou, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - Yixing People's Hospital, Wuxi, Jiangsu
  - The Second Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Fuzhou First People's Hospital of Jiangxi Province, Fuzhou, Jiangxi
  - Nanfang Hospital，Ganzhou, Ganzhou, Jiangxi
  - Jingdezhen No.1 People's Hospital, Jingdezhen, Jiangxi
  - Jiujiang No.1 People's Hospital, Jiujiang, Jiangxi
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - ShangRao People's Hospital, Shangrao, Jiangxi
  - Yugan Xinjiang hospital, Shangrao, Jiangxi
  - Tonggu County People's Hospital, Yichun, Jiangxi
  - Yichun People's Hospital, Yichun, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Anshan Central Hospital, Anshan, Liaoning
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Central Hospital of Wafangdian, Dalian, Liaoning
  - Central Hospital of Zhuanghe City, Dalian, Liaoning
  - Dalian Jinzhou District First People's Hospital, Dalian, Liaoning
  - Dalian Lvshun District Hospitai of tradition Chinese Medicine, Dalian, Liaoning
  - Dalian Lvshun District People's Hospital, Dalian, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Dalian PuLanDian central hospital, Dalian, Liaoning
  - Dalian University Affiliated Xinhua Hospital, Dalian, Liaoning
  - The Second People's Hospital of Huludao, Huludao, Liaoning
  - Panjin Central Hospital, Panjin, Liaoning
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Guyuan people's hospital, Guyuan, Ningxia
  - People's Hospital of Zhongwei, Zhongwei, Ningxia
  - Ankang Central Hospital, Ankang, Shaanxi
  - East District of The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xi 'an Fengcheng Hospital, Xi'an, Shaanxi
  - Xianyang Hospital of Yan 'an University, Xianyang, Shaanxi
  - Zichang People's Hospital, Yan’an, Shaanxi
  - Weihai Wendeng District People's Hospital, Weihai, Shandogn
  - Binzhou Central Hospital, Binzhou, Shandong
  - Yangxin County People Hospital, Binzhou, Shandong
  - Ningjin People's Hospital, Dezhou, Shandong
  - People's Hospital of Qihe County, Dezhou, Shandong
  - The Second People's Hospital of Dongying, Dongying, Shandong
  - Yuncheng County People's Hospital, Heze, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - Liaocheng City Central Hospital, Liaocheng, Shandong
  - Liaocheng People's Hospital（Liaocheng Brain Hospital）, Liaocheng, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The People's Hospital of Gaotang, Liaocheng, Shandong
  - The people's Hospital of Linqing, Liaocheng, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - Third People's Hospital of Liaocheng, Liaocheng, Shandong
  - Yanggu Traditional Chinese Medical Hospital, Liaocheng, Shandong
  - Linyi Central Hospital, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Linyi Third People's Hospital, Linyi, Shandong
  - Linyi Traditional Chinese Medicine Hospital, Linyi, Shandong
  - People's Hospital of Yinan, Linyi, Shandong
  - Qingdao Fuwai Cardiovascular Hospital, Qingdao, Shandong
  - Qixia City People's Hospital, Qixian, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Qixia traditional Chinese medicine hospital, Yantai, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical University, Yantai, Shandong
  - Yantai Penglai People's Hospital, Yantai, Shandong
  - Yantai Penglai traditional Chinese medicine hospital, Yantai, Shandong
  - Yantai Taocun Central Hospital, Yantai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Yantai Zhifu hospital, Yantai, Shandong
  - YEDA hospital, Yantai, Shandong
  - Yicheng Municipal Hospital of Zaozhuang, Zaozhuang, Shandong
  - PKUcare Zibo Hospital, Zibo, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Zibo Hospital of Traditional Chinese Medicine, Zibo, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Shanghai Seventh People's Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Linfen Central Hospital (neurology department), Linfen, Shanxi
  - Linfen Central Hospital(emergency department), Linfen, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First People's Hospital of Longquanyi Disdrict,Chengdu, Chengdu, Sichuan
  - People's Hospital of Deyang City, Deyang, Sichuan
  - The Third Hospital of Mianyang, Mianyang, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Urumqi, China, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Nujiang Lisu Autonomous Prefecture People's Hospital, Nujiang, Yunnan
  - Ninger County People's Hospital, Pu'er, Yunnan
  - Tengchong People's Hospital, Tengyue, Yunnan
  - The First People's Hospital of jiande, Hangzhou, Zhejiang
  - People's Hospital of Anji, Huzhou, Zhejiang
  - Haiyan People's Hospital, Jiaxing, Zhejiang
  - Juancheng County People's Hospital, Heze

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study can be made available to other researchers on reasonable request and after signing appropriate data sharing agreements.

REFERENCES:
- [Derived] Li J, Jing J, Meng X, Shi FD, Gu HQ, Jin A, Jiang Y, Li H, Johnston SC, Hankey GJ, Easton JD, Xie X, Jin WN, Chang L, Shi P, Wang L, Zhuang X, Li H, Zang Y, Zhang J, Sun Z, Liu D, Li Y, Yang H, Zhao J, Yu W, Wang A, Pan Y, Lin J, Li S, Niu S, Wang Y, Zhao X, Li Z, Liu L, Zheng H, Wang Y; CHANCE-3 Investigators. Colchicine for preventing stroke in patients with and without intracranial atherosclerotic stenosis: a prespecified analysis of a randomized clinical trial. EClinicalMedicine. 2025 May 19;84:103226. doi: 10.1016/j.eclinm.2025.103226. eCollection 2025 Jun. PMID 40496882
- [Derived] Li J, Meng X, Shi FD, Jing J, Gu HQ, Jin A, Jiang Y, Li H, Johnston SC, Hankey GJ, Easton JD, Chang L, Shi P, Wang L, Zhuang X, Li H, Zang Y, Zhang J, Sun Z, Liu D, Li Y, Yang H, Zhao J, Yu W, Wang A, Pan Y, Lin J, Xie X, Jin WN, Li S, Niu S, Wang Y, Zhao X, Li Z, Liu L, Zheng H, Wang Y; CHANCE-3 Investigators. Colchicine in patients with acute ischaemic stroke or transient ischaemic attack (CHANCE-3): multicentre, double blind, randomised, placebo controlled trial. BMJ. 2024 Jun 26;385:e079061. doi: 10.1136/bmj-2023-079061. PMID 38925803
- [Derived] Wang Y, Li J, Johnston SC, Hankey GJ, Easton JD, Meng X, Shi FD, Wang Y, Zhao X, Li Z, Liu L, Gu H, Jiang Y, Wang A, Pan Y, Jing J, Niu S, Li H. Colchicine in High-risk Patients with Acute Minor-to-moderate Ischemic Stroke or Transient Ischemic Attack (CHANCE-3): Rationale and design of a multicenter randomized placebo-controlled trial. Int J Stroke. 2023 Aug;18(7):873-878. doi: 10.1177/17474930231172312. Epub 2023 May 11. PMID 37060288